CLINICAL TRIAL: NCT04866108
Title: A Single Center, Open-labeled, Single Arm Phase II Study of Fruquintinib Combined With Capecitabine as First-line Treatment for Advanced Metastatic Colorectal Cancer Unsuitable for Intravenous Chemotherapy
Brief Title: A Phase II Study of Fruquintinib Combined With Capecitabine as First-line Treatment for Advanced Metastatic Colorectal Cancer Unsuitable for Intravenous Chemotherapy
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Beijing Friendship Hospital (Other)
Responsible Party: Principal Investigator, Bai Zhigang, Professor, Beijing Friendship Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HMPL-013-FLAG-C104
Record Dates: First submitted 2021-04-27; First posted 2021-04-29 (Actual); Last update posted 2022-08-18 (Actual); Status verified 2022-08

CONDITIONS: Unresectable Metastatic Colorectal Cancer
MeSH Terms: interventions — HMPL-013; Capecitabine

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental (Experimental): Fruquintinib, 4mg/d, qd po, 2 weeks on, 1 week off; Capecitabine: 825mg/m2, bid po, 2 weeks on, 1 week off
  Interventions: Drug: fruquintinib plus capecitabine

INTERVENTIONS:
Drug: fruquintinib plus capecitabine — oral fruquintinib plus capecitabine

SUMMARY:
This is a single center, open-labeled, single arm phase II study aimed to investigate the efficacy and safety of fruquintinib combined with capecitabine as first-line treatment for advanced metastatic colorectal cancer patients unsuitable for intravenous chemotherapy.

DETAILED DESCRIPTION:
Fruquintinib is an oral small molecule inhibitor of VEGFR1/2/3, this phase II study aimed to investigate the efficacy and safety of fruquintinib combined with capecitabine as first-line treatment for advanced metastatic colorectal cancer patients of elderly or those unsuitable for intravenous chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

1. ≥18 years old at the time of signing the informed consent;
2. Histologically or cytologically confirmed unresectable metastatic colorectal cancer;
3. Haven't received systematic therapy after diagnosis of metastatic colorectal cancer;
4. Intolerable to standard treatment of oxaliplatin- or irinotecan-based intravenous combination therapy;
5. At least one measurable lesion(s);
6. ECOG PS 0-2;
7. Life expectancy≥3 months;
8. Adequate organ and bone marrow functions;
9. Women of childbearing age must have a negative pregnancy test within the first day of the study, and contraceptive methods should be taken during the study until 6 months after the last administration;
10. Willingness and able to comply with scheduled visits, treatment plans, laboratory tests, and other study procedure.

Exclusion Criteria:

1. Previous treatment with VEGFR inhibition;
2. Participating in other drug clinical trials within 4 weeks before recruited;
3. Have received other systemic anti-tumor therapies within 4 weeks before recruited;
4. Non-controlled hypertension after monotherapy, that is, systolic blood pressure > 140mmHg or diastolic blood pressure > 90mmHg;
5. Proteinuria ≥ 2+ (1.0g/24hr);
6. Clinically significant electrolyte abnormality;
7. Clinically significant cardiovascular diseases;
8. Thromboembolism or arteriovenous events occurred 6 months before recruited;
9. ≥grade 3 bleeding events 4 weeks before recruited;
10. Evidence of CNS metastasis;
11. Active gastric and duodenal ulcer, ulcerative colitis or uncontrolled hemorrhage in GI;
12. Active, symptomatic interstitial lung disease causing dyspnea (≥ grade 2 dyspnea), pleural effusion or ascites;
13. History of organ transplantation;
14. APTT >1.5×ULN or INR>1.5;
15. History of HIV infection or active hepatitis B / C;
16. Allergic to fruquintinib and / or capecitabine;
17. Pregnant or lactating women;
18. Clinically detectable secondary primary malignancies at the time of enrollment (excluding fully treated basal cell carcinoma of the skin or carcinoma in situ of the cervix);
19. Patients who are not suitable for the study judged by the researchers.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Estimated)
Dates: Start 2021-12-08 (Actual); Primary Completion 2024-06 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | From Baseline to primary completion date, about 3 years
  ORR according to Response Evaluation Criteria in Solid Tumors (RECIST) version. 1.1

SECONDARY OUTCOMES:
Overall Survival (OS) | From Baseline to primary completion date, about 3 years
  OS is determined from the date of treatment to death from any cause or the last follow-up date
Progression Free Survival (PFS) | From Baseline to primary completion date, about 3 years
  PFS is determined from the date of treatment to PD or death from any cause
Disease Control Rate (DCR) | From Baseline to primary completion date, about 3 years
  DCR according to Response Evaluation Criteria in Solid Tumors (RECIST) version. 1.1
Adverse Events and Serious Adverse Events | From Baseline to primary completion date, about 3 years
  Safety and tolerance will be evaluated by incidence, severity and outcomes of adverse events (AEs) and categorized by severity in accordance with the NCI CTC AE Version 5.0.
Quality of Life (QoL) | From Baseline to primary completion date, about 3 years
  Quality of life is assessed using the European Organization for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire (QLQ) C30. It will be evaluated at Screening, Tumor Assessment Visit and End of Treatment visit.

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Friendship Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wang X, Bai Z, Deng W, Wang X. Efficacy and safety of fruquintinib plus capecitabine as first-line treatment in patients with metastatic colorectal cancer ineligible for intravenous chemotherapy: a two-stage, single-armed, phase II study. Invest New Drugs. 2025 Apr;43(2):214-222. doi: 10.1007/s10637-025-01510-1. Epub 2025 Feb 13. PMID 39945972